CLINICAL TRIAL: NCT06428422
Title: The Impact of Bifidobacterium Lactis Supplementation on Survival and Treatment Response in Metastatic Non-small Cell Lung Cancer Patients Receiving Immunotherapy (Nivolumab)
Brief Title: The Impact of Probiotic on Survival and Treatment Response in Metastatic Non-small Cell Lung Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, Mehmet Artac, Prof.Dr., Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BL-32769
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Non-small Cell Lung Cancer
Keywords: immunotherapy; lung cancer; probiotics; Bifidobacterium animalis; microbiota
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive an oral dosage of 4 x 10^9 cfu/g/day Bifidobacterium animalis subsp. lactis BL-04 strain (Danisco, USA) and 1 gram of maltodextrin (Danisco, USA) in conjunction with the conventional treatment, which consisted of systemic cancer immunotherapy with nivolumab at a dose of 3 mg/kg administered intravenously every two weeks. The immunotherapy with nivolumab will be completed in twelve weeks.
  A probiotic strain is provided to the intervention group in the form of a sachet. Patients will be asked to pour the entire sachet into a glass of water (100 mL, room temperature), mix, and drink it every day for 12 weeks.
  Interventions: Dietary Supplement: Bifidobacterium animalis subsp. lactis Bl-04
- Plasebo group (Placebo Comparator): The plasebo group will receive the conventional treatment, which consisted of systemic cancer immunotherapy with nivolumab at a dose of 3 mg/kg administered intravenously every two weeks. The immunotherapy with nivolumab will be completed in twelve weeks.
  In addition to the traditional treatment (nivolumab), the plasebo group will be given 1 g/day maltodextrin (Danisco, USA) as placebo. Maltodextrin will be provided to the intervention group in the form of a sachet. Patients will be asked to pour the entire sachet into a glass of water (100 mL, room temperature), mix, and drink it every day for 12 weeks.
  Interventions: Other: Plasebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium animalis subsp. lactis Bl-04 — 4 x 10^9 cfu/g/day Bifidobacterium animalis subsp. lactis Bl-04 for 12 weeks
  Arms: Intervention group
Other: Plasebo — 1 g/day maltodextrin for 12 weeks
  Arms: Plasebo group

SUMMARY:
The aim of this study is to evaluate the effect of a probiotic supplement containing Bifidobacterium animalis lactis BL-04 on the clinical effectiveness of immunotherapy in patients diagnosed with metastatic non-small cell lung cancer who are receiving immunotherapy.

DETAILED DESCRIPTION:
Despite modern treatments, lung cancer remains a leading cause of high mortality worldwide. Over the past decade, significant improvements in patient survival have been achieved with immune checkpoint inhibitors, which enhance the T cell-mediated immune response to eradicate cancer cells. However, therapeutic resistance, drug side effects, and heterogeneous treatment responses limit their effectiveness. Recent studies have established a clear relationship between gut microbiota and cancer immunotherapy. The intestinal microbiota has been shown to stimulate the anti-tumor immune response by modulating immune system cells. Evidence from preclinical and clinical studies indicates that gut microbiota plays a crucial role in the efficacy of immunotherapy and the modulation of drug toxicity. Identifying the microbiota as a potential biomarker could facilitate personalized treatment protocols. Genetic, epigenetic, and microbiota modulation factors are essential for optimizing cancer immunotherapy outcomes. Consequently, research is increasingly focusing on personalized treatment protocols for microbiota modulation, including diet regulation, fecal microbiota transfer, prebiotics, and probiotics. There has been a significant rise in studies demonstrating the clinical benefits of microbial therapy products as complementary treatments.

The functional role of microbiota in modulating the systemic immune response has prompted investigations into its impact on cancer immunotherapy, particularly with agents targeting immunological checkpoints like PD-1. Recent studies have identified both positive and negative regulatory bacteria that influence immunotherapy effectiveness. However, sociocultural and dietary lifestyle differences affect gut microbiota composition, leading to variations between populations. Therefore, studies are needed to identify the unique microbiome composition of each population to develop microbiota biological indicators for cancer immunotherapy. No research has been conducted in this area in Türkiye. This study aims to identify bacterial species that may serve as biomarkers for the microbiota specific to Turkish cancer patients receiving immunotherapy and use them for prognostic purposes.

Understanding the significant role of probiotics in modulating intestinal microbiota has increased the demand for these food supplements. Studies show that anti-tumor efficacy is specific to the bacterial strain. For instance, Bifidobacteriums have been reported to enhance the effectiveness of PD-1 blockers in experimental rat models. In another study, B. lactis BL-04 reduced immunotherapy-induced colitis in animals.

This study will investigate the effect of a probiotic supplement containing Bifidobacterium animalis lactis BL-04 on clinical objective response, clinical benefit rates, and intestinal microbiota in patients with metastatic non-small cell lung cancer (mNSCLC) receiving nivolumab. The results may facilitate the development of specific probiotic supplements as a complementary therapy for mNSCLC treatment.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study.
* Histologically confirmed diagnosis of Non-Small Cell Lung Cancer (NSCLC).
* Patients must be in an advanced stage (incurable with surgery or radiotherapy) or have metastatic disease (Stage IV).
* Male or female patients aged >18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status less than 2.
* Laboratory findings must confirm adequate bone marrow function, indicated by:

White Blood Cell (WBC) count > 2,000/mm³, Neutrophil count > 1,500/mm³,Platelet count > 100,000/mm³

Exclusion Criteria:

* Previously received treatment with any of the following antibody blockers: anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4.
* Currently taking probiotic supplements or consuming probiotic bacteria-supported yogurt and similar food supplements.
* Antibiotic utilization within the past month
* Active interstitial lung disease or a history of interstitial lung disease requiring systemic steroid treatment.
* A condition requiring systemic corticosteroids (greater than 10 mg of prednisone daily or equivalent) or who have received immunosuppressive treatment within 14 days prior to the first dose of the study.
* Presence of uncontrolled adrenal insufficiency.
* Pregnancy or breastfeeding.
* Severe congestive heart failure (Class III or higher according to the New York Heart Association Functional Classification) or a history of myocarditis.
* Uncontrolled cardiac arrhythmia that developed within six months prior to the start of the study.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Clinical Response | Week 12
  The clinical impact of the immunotherapy will be evaluated according to RECIST (Response Evaluation Criteria In Solid Tumors) 1.1 criteria based on radiological analysis.
Progression-free survival | Basaline and the date of radiological progression
  The progression-free survival (PFS) period will be defined as the interval between the initiation of treatment and the date of radiological progression.
Overall survival | Basaline and the date of death from any case
  The overall survival (OS) period will be defined as the interval between the date of disease diagnosis and death from any cause.

SECONDARY OUTCOMES:
Intestinal microbiota modulation | Basaline and Week 12
  Microbiota and fatty acid analyses, including acetic acid, propionic acid, and butyric acid, will be conducted on fecal samples."
Immunological findings | Basaline and Week 12
  The concentrations of CD4+ T cell subgroups (Th1, Th2, Th9, Th17, Th1Th17, and Treg) and sitokins (IL-1β, IL-4, IL-10, IL-17, TNF-α, TGF-beta, IFN-gamma, IL-36 and trimethylamine N-oxide) will be quantified in the serum samples of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No